CLINICAL TRIAL: NCT05328869
Title: The Effects Of Relaxation Training In Women With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/04/07
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation group (Experimental): Jacobson progressive relaxation training will be applied
  Interventions: Other: Relaxation training
- Control group (Other): No intervention will be applied
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Relaxation training — Relaxation training will be performed under the supervision of a physiotherapist. The training is carried out from the estimated day of ovulation (cycle length in days minus 14) until the next menstrual period begins
  Arms: Relaxation group
Other: No intervention — No intervention will be applied. The natural process will be followed from the estimated day of ovulation (cycle length in days minus 14) until the next menstrual period begins
  Arms: Control group

SUMMARY:
The aim of this study was to investigate the effects of relaxation training on menstrual pain severity, menstrual symptoms, impact of quality of life, impact of work/academic performance, impact of social activity level and anxiety level in women with primary dysmenorrhea (PD) complaints.

DETAILED DESCRIPTION:
PD is the cramping pain that comes before or during a menstrual period. Relaxation training contributes to the reduction of stress and pain. Thus, there is a need to investigate the effects of relaxation training in dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary dysmenorrhea complaint according to the Primary Dysmenorrhea Consensus Guide,
* Over 18 years of age,
* Having a mean pain intensity of moderate and higher according to the Visual Analogue Scale in the last 6 months,
* Having a regular menstrual cycle (28±7 days),
* Volunteered to participate in the study.

Exclusion Criteria:

* Having a pathological history and radiological findings pointing to secondary dysmenorrhea,
* Using oral contraceptives/antidepressants at least 6 months,
* Receiving hormone therapy,
* Undergoing pelvic surgery,
* Pregnant,
* Giving birth,
* Using an intrauterine device,
* Having neurological, orthopedic and/or rheumatological diseases
* Having a psychiatric disease,
* Having a history of malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Primary dysmenorrhea is a gynecological problem that can be seen in most women.
Enrollment: 30 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Menstrual pain intensity | change from baseline at an average of 2 weeks
  Menstrual pain intensity will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "no pain", while "10" = "unbearable pain". Individuals will be asked to mark on a 10 cm straight line according to the level of pain they feel. Pain intensity will be recorded by measuring the distance between the beginning of the line and the marked place.

SECONDARY OUTCOMES:
Menstrual symptoms | change from baseline at an average of 2 weeks
  Menstrual symptoms will be measured with the menstrual symptom questionnaire. Menstrual Symptom Questionnaire is a 24-item self-report scale and each item is scored between 1 (never) and 5 (always). An increase in the mean score indicates an increase in the severity of menstrual symptoms. The total score is 120 points.
Impacts of academic/work performance | change from baseline at an average of 2 weeks
  Impacts of academic/work performance will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0"= means "my work/school performance is not affected in any way", while "10"= means "my work/school performance is greatly affected"
Impacts of life quality | change from baseline at an average of 2 weeks
  Impacts of life quality will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "my quality of life is not affected in any way", while "10" = "my quality of life is greatly affected". Individuals will be asked to mark on a 10 cm straight line according to the quality of life they think.
Impacts of social activity | change from baseline at an average of 2 weeks
  Impacts of social activity will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "my social activity is not affected in any way", while "10" = "my social activity is greatly affected". Individuals will be asked to mark on a 10 cm straight line according to the social activity they think.
Anxiety level | change from baseline at an average of 2 weeks
  Anxiety level will be assessed with the Spielberger State Trait Anxiety Inventory. This inventory is a 40-item self-report inventory designed to measure both state anxiety section (current feelings of apprehension, worry, etc.) and trait anxiety section (continuous feelings of apprehension, worry, etc.). Each section is scored on four levels of anxiety intensity from 1="not at all" to 4="very much" and with a sum score between 20 and 80. A higher total score indicates more severe anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University